CLINICAL TRIAL: NCT01071278
Title: Lipid Management in Clinical Practice
Brief Title: Lipid Management in Clinical Practice (MK-0524A-115)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0524A-115; 2010_011 (Other: Merck Study Number)
Record Dates: First submitted 2010-02-17; First posted 2010-02-19 (Estimated); Results first posted 2012-03-07 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-07

CONDITIONS: Lipid Metabolism Disorder
Keywords: Lipid metabolism disorder
MeSH Terms: conditions — Lipid Metabolism Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients treated within a disease management program: Participant prescribed Tredaptive® for dyslipidemia and also participated in a disease management program for treatment of diabetes mellitus, coronary heart disease or both.
- Patients treated outside a disease management program: Participant prescribed Tredaptive® for dyslipidemia and did not participate in a disease management program for treatment of diabetes mellitus, coronary heart disease or both.

SUMMARY:
The aim of this observational program is to generate data on the use of Tredaptive (nicotinic acid/laropiprant) for lipid management under routine medical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients are 18 years of age or older with lipid disorder treated with nicotinic acid/laropiprant

Exclusion Criteria:

* Patient is currently participating in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in routine medical care either statutorily health insured or privately insured
Sampling Method: Probability Sample
Enrollment: 2390 (Actual)
Dates: Start 2009-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- All Evaluable Participants: Participants who were prescribed Tredaptive® for the treatment of dyslipidemia and primary hypercholesterolemia as per the Summary of Product Characteristics (SmPC) by his/her primary physician in a routine clinical setting either within or outside a Disease Management Program (DMP).
Period: Overall Study
Arm/Group | All Evaluable Participants
Started | 2390
Completed | 1677
Not Completed | 713
Not completed — Premature Discontinuation | 254
Not completed — Completion Status Unknown | 459

BASELINE CHARACTERISTICS:
Groups:
- Intent-to-Treat Population: Baseline characteristics were reported for the 2359 participants in the Intent-to-Treat (ITT) Population, which included all participants from the Evaluable Population who began therapy at or after Visit 1. The ITT Population excluded 31 of the 2390 evaluable participants who began treatment prior to Visit 1.
Arm/Group | Intent-to-Treat Population
Number analyzed (Participants) | 2359
Age, Continuous [Mean (Full Range); unit: years] — Age data was missing 13 of the 2359 participants in the ITT Population.
  years | 61.1 [20 to 94]
Sex/Gender, Customized [Number; unit: participants]
  Male | 1572
  Female | 776
  Not reported | 11
Region of Enrollment [Number; unit: participants]
  Germany | 2359

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Lipid Panel Control
Description: Lipid Panel Control was defined as achieving target for one or more of the following parameters: low-density lipoprotein cholesterol (LDL-C) at goal (<100mg/dL), high-density lipoprotein cholesterol (HDL-C) within normal range (40mg/dL for males and 50mg/dL for females), and/or triglycerides within normal range (≤ 150mg/dL).
Time Frame: From Visit 1 entrance evaluation (Week 0) to Visit 2 (between Weeks 8-22)
Population: Results are for the Intent-to-Treat (ITT) Population. Information regarding the participation in a disease management program was not reported for 63 participants in the ITT Population.
Measure: Number; unit: participants
Arm/Group | Patients Treated Within a Disease Management Program | Patients Treated Outside a Disease Management Program
Number analyzed (Participants) | 1224 | 1072
participants
  1 lipid parameter | 249 | 192
  2 lipid parameters | 245 | 231
  3 lipid parameters | 232 | 194
  No lipid parameter | 70 | 33
  Not Reported | 428 | 422

2. Secondary Outcome: Number of Participants Who Reported Adverse Events
Time Frame: Up to 22 weeks
Measure: Number; unit: participants
Arm/Group | All Evaluable Participants
Number analyzed (Participants) | 2390
participants
  Leukocytosis | 1
  Acute Myocardial Infarction | 1
  Angina Pectoris | 1
  Cardiovascular Disorder | 1
  Coronary Artery Insufficiency | 1
  Tachycardia | 3
  Eyelid Oedema | 1
  Visual Impairment | 2
  Abdominal Discomfort | 7
  Abdominal Distension | 1
  Abdominal Pain | 3
  Abdominal Pain Upper | 9
  Constipation | 1
  Diarrhoea | 13
  Dyspepsia | 4
  Eructation | 1
  Flatulence | 3
  Gastrointestinal Disorder | 1
  Irritable Bowel Syndrome | 1
  Lip Swelling | 1
  Nausea | 30
  Pancreatic Cyst | 1
  Pancreatitis Chronic | 1
  Vomiting | 9
  Adverse Event | 4
  Asthenia | 1
  Chills | 2
  Condition Aggravated | 1
  Drug Ineffective | 6
  Drug Intolerance | 1
  Face Oedema | 1
  Fatigue | 2
  Feeling Abnormal | 1
  Feeling Hot | 9
  Hyperthermia | 1
  Malaise | 4
  Oedema | 1
  Oedema Peripheral | 2
  Pain | 2
  Swelling | 1
  Cholelithiasis | 1
  Hypersensitivity | 3
  Diverticulitis | 1
  Gastroenteritis | 1
  Rash Pustular | 1
  Splenic Abscess | 1
  Accident | 1
  Alanine Aminotransferase Increased | 1
  Blood Cholesterol Abnormal | 2
  Blood Cholesterol Increased | 1
  Blood Creatine Phosphokinase Increased | 1
  Blood Creatinine Increased | 3
  Blood Glucose Abnormal | 1
  Blood Glucose Fluctuation | 1
  Blood Glucose Increased | 5
  Blood Pressure Decreased | 1
  Blood Triglycerides Abnormal | 2
  Blood Triglycerides Increased | 5
  Blood Uric Acid Increased | 1
  Gamma-Glutamyltransferase Increased | 2
  Lipids Abnormal | 1
  Lipids Increased | 1
  Lipoprotein (A) Increased | 1
  Weight Increased | 1
  Diabetes Mellitus | 2
  Diabetes Mellitus Inadequate Control | 1
  Gout | 2
  Hyperglycaemia | 1
  Lactose Intolerance | 1
  Lipid Metabolism Disorder | 1
  Arthralgia | 1
  Muscular Weakness | 1
  Musculoskeletal Discomfort | 1
  Musculoskeletal Stiffness | 1
  Myalgia | 6
  Pain In Extremity | 1
  Spondylitis | 1
  Multiple Myeloma | 1
  Burning Sensation | 4
  Dizziness | 10
  Dysaesthesia | 1
  Headache | 9
  Hypotonia | 1
  Paraesthesia | 10
  Anxiety | 3
  Depressed Mood | 1
  Depression | 1
  Fear | 1
  Insomnia | 1
  Loss of Libido | 1
  Restlessness | 7
  Sleep Disorder | 1
  Asthma | 1
  Dyspnoea | 4
  Increased Upper Airway Secretion | 1
  Cold Sweat | 1
  Dermatitis Allergic | 1
  Eczema | 4
  Erythema | 17
  Hyperhidrosis | 3
  Petechiae | 1
  Pruritus | 31
  Pruritus Generalised | 7
  Rash | 9
  Skin Burning Sensation | 3
  Skin Disorder | 1
  Skin Reaction | 1
  Skin Swelling | 1
  Swelling Face | 2
  Urticaria | 4
  Appendicectomy | 1
  Pain Management | 1
  Vascular Graft | 1
  Flushing | 54
  Hot Flush | 8
  Hypertension | 1

ADVERSE EVENTS:
Arm/Group | All Evaluable Participants
Serious Adverse Events (participants affected / at risk) | 20/2390
Other Adverse Events (participants affected / at risk) | 0/2390
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Evaluable Participants (N=2390)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Coronary Artery Insufficiency (Cardiac disorders) | 1 (1)
Lip Swelling (Gastrointestinal disorders) | 1 (1)
Pancreatic Cyst (Gastrointestinal disorders) | 1 (1)
Pancreatitis Chronic (Gastrointestinal disorders) | 1 (1)
Feeling Hot (General disorders) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Splenic Abscess (Infections and infestations) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1)
Blood Cholesterol Abnormal (Investigations) | 1 (1)
Blood Creatinine Increased (Investigations) | 2 (2)
Blood Triglycerides Abnormal (Investigations) | 2 (2)
Blood Triglycerides Increased (Investigations) | 1 (1)
Lipoprotein (A) Increased (Investigations) | 1 (1)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 (1)
Lipid Metabolism Disorder (Metabolism and nutrition disorders) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Swelling Face (Skin and subcutaneous tissue disorders) | 1 (1)
Appendicectomy (Surgical and medical procedures) | 1 (1)
Pain Management (Surgical and medical procedures) | 1 (1)
Skin Swelling (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MSD SHARP & DOHME GmbH and its comarketing companies have exclusive rights to the use and evaluation of the data collected in this study.